CLINICAL TRIAL: NCT07377630
Title: Intrathecal MoRphine Versus Transabdominal Plane Block (TAP) Block for AnalGesic Management in Elective Caesarean Section Performed Under Neuraxial Anesthesia. A Monocentric Pilot Randomized Controlled Trial
Brief Title: Intrathecal MoRphine Versus Transabdominal Plane Block (TAP) Block for AnalGesic Management in Elective Caesarean Section
Acronym: MIRAGE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EU CT 2024-513150-29-00
Record Dates: First submitted 2025-08-07; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Cesarean Section; Neuroaxial Analgesia Procedures
Keywords: cesarean section; neuraxial anesthesia; TAP block; morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal morphine as adjuvant (ITM group) (Experimental): All patients will undergo spinal anesthesia at the L3 to L4 or L4 to L5 interspace with hyperbaric bupivacaine 0.5% (10 mg) and 3 μg of sufentanil, Intrathecal morphine as adjuvant (ITM) group adds morphine 30 μg.
  Interventions: Drug: Intrathecal Morphine
- TAP block with ropivacaine and clonidine (TB) (Active Comparator): At the end of surgery, in the TB group a bilateral ultrasound-guided Transabdominal Plane Block (TAP) block is performed with 20 ml of ropivacaine 0.25% and 75 μg of clonidine each site using a non-Insulated Echogenic Needle 22 Gauge (80 mm). The TAP block will be performed behind the operating drapes so the patient remains blind to the study arm.
  Interventions: Drug: TAP Block

INTERVENTIONS:
Drug: Intrathecal Morphine — The anesthetist in charge performs spinal anesthesia using a 25-gauge pencil point needle in the sitting position at the L3 to L4 or L4 to L5 interspace. After skin disinfection with 2% alcoholic chlorhexidine solution and skin anesthesia with 2 ml of lidocaine 2%, all patients receive spinal anesthesia with a solution of 2 ml hyper-baric bupivacaine 0.5% (10 mg) and 3 μg of sufentanil while, ITM group adds morphine 30 μg. The patient is not informed about the drugs used in spinal anesthesia.
  Arms: Intrathecal morphine as adjuvant (ITM group)
Drug: TAP Block — At the end of surgery, in the TB group a bilateral Transabdominal Plane Block (TAP) block is performed. The anesthetist prepares two sy-ringes with 20 ml each with ropivacaine 0.25% with 75 μg of clonidine. Upon identifying the TAP compart-ment in the lateral abdominal wall (in the midaxillary line between the bony prominences of the subcostal margin and the iliac crest) with the linear high-frequency ultrasound probe, we penetrate the skin with the block needle using an in-plane technique. Upon entering the plane between the internal oblique and the transversus abdominis muscles, and after negative aspiration of blood, the local anesthetic is slowly injected. The TAP compartment begins to separate, hydrodissect, or "unzip" as the local anesthetic is injected, pushing the transversus abdominis muscle down. An injection of 20 ml of the prepared solution is injected for each side. The TAP block is performed behind the operating drape.
  Arms: TAP block with ropivacaine and clonidine (TB)

SUMMARY:
The goal of this randomized controlled clinical trial is to determine if low-dose intrathecal morphine is superior to a Transversus Abdominis Plane (TAP) block with ropivacaine and clonidine for postoperative analgesia in women aged 18 years or older undergoing elective cesarean section under neuraxial anesthesia.

The main questions it aims to answer are:

* Is intrathecal morphine more effective than TAP block in reducing postoperative somatic pain at rest?
* Does intrathecal morphine differ from TAP block in terms of adverse events, pain during mobilization, visceral pain, rescue analgesic use, maternal satisfaction, and newborn wellbeing?

Researchers will compare the intrathecal morphine (ITM) group to the TAP block (TB) group to see if ITM provides superior analgesia and improved secondary outcomes.

Participants will:

* Undergo spinal anesthesia with hyperbaric bupivacaine and sufentanil
* add 30 μg intrathecal morphine (only ITM group)
* receive bilateral ultrasound-guided TAP block with 20 ml ropivacaine 0.25% and 75 μg clonidine per side (only TB group)
* receive standardized postoperative analgesia with paracetamol, ibuprofen, and tramadol as needed
* be monitored postoperatively for pain (somatic and visceral, at rest and with movement), adverse events, mobilization, maternal satisfaction, and newborn outcomes at regular intervals for 24 hours

This is a single-center, pilot, single-blind trial involving 100 participants (50 per group).

DETAILED DESCRIPTION:
It is a monocentric randomized single-blind controlled pilot trial, wherein the patient and the biostatistics will be unaware about assigned treatment group, whereas the study investigators and site staff will be aware of the treatment group.

The trial consists in two treatment arms:

* Transabdominal Plane Block (TAP) block with ropivacaine and clonidine performed at the end of surgery (this will be performed in the operating room, behind a drape, so that the patient is unaware of the study arm)
* Addition of low doses of morphine to the other drugs administered during the performance of spinal anaesthesia Women aged 18 years and older, with indication for elective caesarean section, gestational age 34 weeks and older, admitted to the Giannina Gaslini Institute will participate in this study.

After an adequate anamnesis, the confirmation of the presence of all the inclusion criteria and the absence of the exclusion criteria and the acquisition of the informed consent, the subjects will be assigned to the treatment arm with a computer-generated random number sequence. The investigator/designated study personnel will administer the treatment as per the randomization codes.

Clinical and instrumental parameters (such as pain, vital signs, the possible occurrence of symptoms such as nausea, vomiting, itching) will then be evaluated during the caesarean section and at 12, 18, 24 hours on the day of the caesarean section (possibly at 6 a.m. on the following day in the case of a caesarean section after 12 noon) and 24 hours after the operation, and the use of analgesics as needed in the case of uncontrolled pain (previously prescribed by the anaesthetist). The baby's well-being will be assessed at birth and, 24 hours after the operation, a questionnaire will be submitted to the patient, to assess her satisfaction.

The study intervention will be performed in the operating room of Departmental Unit of Obstetrics and Gyne-cology of IRCSS Giannina Gaslini Institute. The follow up will be performed in the inpatient ward of the same Departmental Unit.

For the purpose of this trial, the end of study (EOS) is defined as the last visit of last patient.

A total number of 100 participants, a sample size of 50 per group, will be recruited during the study.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective Cesarean Section (CS)
* Scheduled for spinal anesthesia
* Gestational age > 34 weeks
* Age 18 years or above
* Ability to read and understand the information sheet and to sign and date the consent form

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification >2
* Body Mass Index (BMI) ≥ 40 kg/m2
* Weight < 50 kg
* Height < 150 cm or ≥ 180 cm
* Complicated Pregnancy (abnormal placentation, preeclampsia or others)
* Women with opioid use disorder
* Contraindication to spinal anesthesia (clotting disorder, local infection, spinal malformation, elevated intracranial pressure)
* Contraindication to Transabdominal Plane Block (TAP) block (skin infection, abdominal wall muscle defects)
* Allergy/contraindication to any medication used in the study
* Previous median abdominal incision
* Emergency or unplanned CS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
The primary object is to determine if, in elective cesarean section performed under neuraxial anesthesia, low dose morphine as intrathecal adjuvant is superior to TAP Block using ropivacaine and clonidine in terms of postoperative pain | From enrollment to 24 hours after spinal anesthesia
  The primary endpoint of this trial is the determination of how many times somatic Visual Analogue Scale (or VAS, from worst 0 to best 10) at rest is 6 or more in the different evaluations at 12 AM, 6 PM, 00 AM (or at 6 PM, 00 AM and 6 AM if the cesarean section is performed after 12 AM) and at 24 hours from the spinal anesthesia.

SECONDARY OUTCOMES:
Evaluation of somatic pain with movement | From enrollment to 24 hours after spinal anesthesia
  STATISTICAL DIFFERENCE OF MEAN AND STANDARD DEVIATION (SD) OF Somatic Pain (with visual analogue scale 0 worst-10 best)
Evaluation of visceral pain at rest and on movement | From enrollment to 24 hours after spinal anesthesia
  STATISTICAL DIFFERENCE OF MEAN AND STANDARD DEVIATION (SD) of Visceral Pain (with visual analogue scale 0 worst-10 best)
Evaluation of rescue dose therapy consumption in mg | From enrollment to 24 hours after spinal anesthesia
  STATISTICAL DIFFERENCE OF MEAN AND STANDARD DEVIATION OF Time to First Rescue Dose (min)
Incidence of adverse events | From enrollment to 24 hours after spinal anesthesia
  Measure the incidence of Nausea (Internal Gaslini scale, 0 best - 4 worst), incidence of pruritus (Internal Gaslini scale, 0 best - 3 worst), incidence of Urinary Retention (occurrence and need for catheterization), incidence of Hypothension (systolic arterial pressure <100 mmHg or <80% of baseline, total mg of ephedrine) and Bradycardia (heart rate <50 bpm)
Evaluate the quality of recovery after surgery for cesarean delivery | From enrollment to 24 hours after spinal anesthesia
  MEAN AND STANDARD DEVIATION OF Obstetric Quality-of-Recovery score ObsQoR-11 (worst 0-best110 pts)
Incidence of Hypotension | From enrollment to 24 hours after spinal anesthesia
  Measurement thorugh systolic arterial pressure <100 mmHg or <80% of baseline, total mg of ephedrine and evaluation of Bradycardia as heart rate <50 bpm

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No